CLINICAL TRIAL: NCT07039760
Title: An Early Phase 1 Study of Asciminib With or Without Sildenafil for Brain Tumors
Brief Title: Asciminib With or Without Sildenafil for Brain Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202509139
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Brain Tumor
Keywords: Asciminib; Sildenafil; ABL1; ABL2; Tyrosine kinase inhibitor; Pediatric brain tumor; Brain tumor; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Brain Neoplasms | interventions — asciminib; Sildenafil Citrate; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Asciminib (Experimental): Patients will receive 1.3 mg/kg oral asciminib 12 +/- 1.5 hours prior to a second dose of 1.3 mg/kg oral asciminib. Surgery or biopsy will take place 3 +/- 1.5 hours after last dose.
  Interventions: Drug: Asciminib; Procedure: Surgical resection or biopsy
- Group B: Asciminib + Sildenafil (Experimental): Patients will receive 1.3 mg/kg oral asciminib plus 20 mg sildenafil (10 mg if < 20 kg) 12 +/- 1.5 hours prior to a second dose of 1/3 mg/kg asciminib plus 20 mg (10 mg if < 20 kg) sildenafil. Surgery or biopsy will take place 3 +/- 1.5 hours after last dose.
  Interventions: Drug: Asciminib; Drug: Sildenafil; Procedure: Surgical resection or biopsy

INTERVENTIONS:
Drug: Asciminib — Commercially available stock
Drug: Sildenafil — Commercially available stock
  Arms: Group B: Asciminib + Sildenafil
Procedure: Surgical resection or biopsy — Standard of care

SUMMARY:
Dissemination of medulloblastoma is an independent risk factor of poor prognosis. Dissemination of medulloblastoma at recurrence is nearly universally fatal. ABL1 and 2 have been recently found to mediate the dissemination of medulloblastoma. Genetically inactivating ABL1 and 2 resulted in decreased leptomeningeal medulloblastoma and improved overall survival (OS) in rodent models. Asciminib is an FDA approved for the treatment of chronic myeloid leukemia and is well tolerated, likely due to its specificity for ABL1 and ABL2. Asciminib is a P-glycoprotein (P-gp) substrate and thus may be susceptible to being pumped out of tumor cells and brain endothelial cells. It is unclear if asciminib can enter the central nervous system (CNS) and brain tumors in adequate concentration to have anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-25 years old, inclusive.
* Radiographic evidence of a recurrent/progressive brain tumor.
* Tumor must be predominantly in an intraparenchymal location.
* Deemed operable (able to be resected or have an open or stereotactic needle biopsy) by treating neurosurgeon.
* Karnofsky/Lansky Performance Status of ≥ 60. Patients who are unable to walk because of paralysis but who are up in a wheelchair will be considered ambulatory for the purposes of the performance score.
* Bone Marrow:

  * ANC (Absolute neutrophil count) ≥ 1000/µl (unsupported).
  * Platelets ≥ 100,000/µl (may be supported by transfusion).
  * Hemoglobin > 8 g/dL (may be supported by transfusion).
* Renal:

  * Serum creatinine ≤ upper limit of institutional normal.
* Hepatic:

  * Bilirubin ≤ 1.5 times upper limit of normal for age.
  * ALT (SGPT) ≤ 3 times institutional upper limit of normal for age.
  * AST (SGOT) ≤ 3 times institutional upper limit of normal for age.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants. All patients and/or their parents or legal guardians must sign an IRB approved written informed consent document.

Exclusion Criteria:

* Tumors suspected to be pituitary tumors or tumors of the meninges.
* Diagnosis of atypical teratoid rhabdoid tumor (ATRT) or diagnosis of pilocytic astrocytoma (PA).
* Unable to take tablets orally
* Pregnant and/or breastfeeding. Subjects of childbearing potential must have a negative serum or urine pregnancy test within 10 days prior to Day 1.
* Active infection requiring treatment or an unexplained febrile (> 101.5o F) illness.
* Known immunosuppressive disease or human immunodeficiency virus infection.
* Any active renal, cardiac (congestive cardiac failure, myocardial infarction, myocarditis), or pulmonary disease.
* Any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction).
* Inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Tumor:plasma ratio of asciminib | At time of surgical resection or biopsy (day 1)
Tumor:plasma ratio of asciminib with sildenafil | At time of surgical resection or biopsy (day 1)

SECONDARY OUTCOMES:
Change in plasma levels of asciminib | Baseline, time of tumor resection/biopsy (day 1), and 8 (+/- 4 hours) after surgical resection or biopsy
Expression of c-MYC in brain tumor specimens | At time of surgical resection or biopsy (day 1)
Expression of p-CRKL in brain tumor specimens | At time of surgical resection or biopsy (day 1)
Proportion of patients with unacceptable toxicity | From start of treatment (day 1) through 3 weeks following asciminib

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thompson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu